CLINICAL TRIAL: NCT02972450
Title: A Phase I/II Randomised Therapeutic HIV Vaccine Trial in Individuals Who Started Antiretrovirals During Primary or Chronic Infection
Brief Title: An HIV Vaccine Trial in Individuals Who Started ART During Primary or Chronic Infection
Acronym: EHVAT01
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Due to the bankruptcy of FITBiotech, the provider of the GTU DNA vaccine.
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Collaborators: European Commission (Other); Swiss Government (Unknown); Medical Research Council (Other Government); FIT Biotech Ltd. (Unknown); Fred Hutchinson Cancer Center (Other); University College, London (Other); Centre Hospitalier Universitaire Vaudois (Other); Imperial College London (Other); Istituto Nazionale per le Malattie Infettive "Lazzaro Spallanzani" IRCCS (Network); Universitätsklinikum Hamburg-Eppendorf (Other); Institut d'Investigacions Biomèdiques August Pi i Sunyer (Other); Henri Mondor University Hospital (Other); European Georges Pompidou Hospital (Other); Saint-Louis Hospital, Paris, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EHVA T01/ANRS VRI05
Record Dates: First submitted 2016-11-10; First posted 2016-11-23 (Estimated); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: HIV-1-infection
MeSH Terms: interventions — vedolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Injection only: Active:placebo (3:1) (Experimental): GTU-MultiHIV B-clade + MVA HIV-B:
  GTU-MultiHIV B-clade - 2 mg of DNA in 1ml encoding a multi HIV antigen (synthetic fusion protein) administered intramuscularly into the non-dominant deltoid muscle at weeks 0 and 4 and MVA HIV-B 0.5ml(1 x108 pfu/ml) MVA encoding the full-length codon-optimized sequence of Gag administered intramuscularly into the non-dominant deltoid muscle at week 12.
  Interventions: Biological: GTU-MultiHIV B-clade vaccine + MVA HIV-B HIV vaccine; Biological: GTU-MultiHIV B-clade vaccine + MVA HIV-B HIV vaccine+ Vedolizumab
- Infusion only: Active:placebo (3:1) (Experimental): Vedolizumab will be administered in the participant's dominant arm as an intravenous infusion over 30 mins.
  Interventions: Drug: Vedolizumab 300 MG [Entyvio]
- Injection and Infusion: Active:placebo (3:1) (Experimental): GTU-MultiHIV B-clade + MVA HIV-B + Vedolizumab
  Interventions: Biological: GTU-MultiHIV B-clade vaccine + MVA HIV-B HIV vaccine; Biological: GTU-MultiHIV B-clade vaccine + MVA HIV-B HIV vaccine+ Vedolizumab; Drug: Vedolizumab 300 MG [Entyvio]
- Placebo (Placebo Comparator): Placebo1 for DNA: Sodium chloride for injection, 0.9% in 1ml administered intramuscularly into the non-dominant deltoid muscle at weeks 0 and 4.
  Placebo 2 for MVA: S08 buffer in 0.5ml administered intramuscularly into the non-dominant deltoid muscle at week 12.
  Placebo for mAb: Sodium Chloride (NaCl) for infusion, 0.9% in 250 ml infusion bags.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GTU-MultiHIV B-clade vaccine + MVA HIV-B HIV vaccine — The vaccine is a solution of HIV MVA vectors (see section 1.3.2) in S08 buffer (10mM Tris/hydrochloride (Tris/HCl), Saccharose 5% (w/v), 10mM Sodium Glutamate (Na Glu), 50mM Sodium Chloride (NaCl), water PPI, pH 8.0).
  0.5ml of ANRS MVA HIV-B (1 x 108 pfu/ml) or placebo for MVA (S8 buffer) will be administered intramuscularly in the deltoid muscle of the non-dominant upper arm. Participants will be observed for one hour after the injection.
  Arms: Injection and Infusion: Active:placebo (3:1); Injection only: Active:placebo (3:1)
Biological: GTU-MultiHIV B-clade vaccine + MVA HIV-B HIV vaccine+ Vedolizumab — The vaccine is a solution of HIV MVA vectors (see section 1.3.2) in S08 buffer (10mM Tris/hydrochloride (Tris/HCl), Saccharose 5% (w/v), 10mM Sodium Glutamate (Na Glu), 50mM Sodium Chloride (NaCl), water PPI, pH 8.0).
  0.5ml of ANRS MVA HIV-B (1 x 108 pfu/ml) or placebo for MVA (S8 buffer) will be administered intramuscularly in the deltoid muscle of the non-dominant upper arm. Participants will be observed for one hour after the injection. Vedolizumab is administered as an intravenous infusion over 30 mins in the dominant arm. After infusion, the line should be flushed with 30mls of normal saline.
  Arms: Injection and Infusion: Active:placebo (3:1); Injection only: Active:placebo (3:1)
Drug: Vedolizumab 300 MG [Entyvio] — Vedolizumab is administered as an intravenous infusion over 30 mins in the dominant arm. After infusion, the line should be flushed with 30mls of normal saline.
  Arms: Infusion only: Active:placebo (3:1); Injection and Infusion: Active:placebo (3:1)
Other: Placebo — Placebo for MVA it is a solution composed of S08 buffer (as for the MVA vaccine) that will be administered intramuscularly in the deltoid muscle of the non-dominant upper arm. Participants will be observed for one hour after the injection.
  Placebo for GTU-MultiHIV B-clade vaccine: Sodium Chloride (NaCl) for infusion, 0.9%.
  Placebo for Vedolizumab: Sodium Chloride (NaCl) for infusion, 0.9% in 250 ml infusion bags.
  Arms: Placebo

SUMMARY:
EVHA T01 is an international, phase I/II, multicentre, multi-stage, double-blind study that will evaluate at least three experimental arms compared to placebo control in HIV-1 infected participants to see if one or more has a clinically relevant impact on the control of viral replication.

DETAILED DESCRIPTION:
The randomization ratio is 1:1:1:1 for vaccine: vedolizumab: combination: placebo in one of 3 schedules.

The study contains a phase I component in order to evaluate the local and systemic reactogenicity following the first administration of products in the first 12 participants. The phase I will consist of a slow enrolment of the first 12 participants who will be randomised at a maximum rate of 1 per week for 4 weeks, then 2 per week for 4 weeks before increasing to 4 or more per week. The IDMC will review of cumulative adverse event data through to and including the first safety visit in the 12th participant and their recommendation will be sought with regard to expanding recruitment.

The phase II component will assess the effectiveness and safety of the three experimental strategies upon viral control following analytic treatment interruption (ATI). The phase II component is divided into two stages, an interim efficacy stage and a final efficacy stage. There will be a pause in enrolment after 88 participants have been enrolled. A planned interim review by the IDMC at the end of the first stage will provide an opportunity to modify the design of subsequent stages or the recruitment strategy.

Screening will take place during the 6 weeks prior to randomisation. Eligible participants will be enrolled at week 0 and randomised to vaccine, vedolizumab, the combination of vaccine and vedolizumab or matched placebos. Participants and study staff will be aware of the schedule the participant is randomised to, with a third allocated to injections, a third to infusions and a third to the combination of injections and infusions. Only staff authorised to prepare the products will know who is randomised to active product or placebo within each schedule in a ratio of 3:1 respectively.

The vaccine regimen will start at week 0 and the vedolizumab regimen at week 2, each with matched placebo.

Participants will continue on cART during the first 24 weeks covering the vaccination period and 5 of 6 vedolizumab/placebo infusions.

Treatment will then be interrupted and resumed when the viral load is confirmed to have rebounded to ≥10,000 copies/ml, or the CD4 falls to ≤350 cells/mm3, or there is evidence of disease progression, or they have completed 24 weeks of treatment interruption.

ELIGIBILITY:
Inclusion Criteria

1. HIV-1-infected
2. Aged 18 - 65 years old on the day of screening
3. Weight >50kg
4. Willing and able to provide written informed consent
5. Nadir CD4 count > 300 cells/mm3
6. CD4 count at screening > 500 cells/mm3
7. Viral load <50 copies/ml at screening
8. Started cART after 2009 and on cART for at least one year prior to screening
9. Willing to interrupt cART for up to 24weeks and change cART regimen if required
10. If sexually active, willing to use a reliable method of reducing the risk of transmission to their sexual partners during treatment interruption (which could include PrEP for their sexual partners)
11. If heterosexually active and able to have children, willing to use a highly effective method of contraception with partner (combined oral contraceptive pill; injectable or implanted contraceptive; IUD/IUS; physiological or anatomical sterility (in self or partner) from 2 weeks before enrolment until 18 weeks after the last injection/infusion
12. If women of childbearing potential*, willing to undergo urine pregnancy tests prior to administration of an injection or an infusion
13. Willing to avoid all other vaccines within 4 weeks of scheduled study injections
14. Willing and able to comply with visit schedule and provide blood samples
15. Being covered by medical insurance or in National Healthcare System

    * A woman will be considered of childbearing potential following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy.

Exclusion criteria:

1. Pregnant or lactating
2. HIV-2 infection (either isolated or associated with HIV-1)
3. VL >200 copies/ml on 2 occasions in the 12 months prior to screening
4. Previous interruptions in cART
5. Previous virological failures defined by loss of virological suppression with the presence of resistant mutations
6. Haemoglobin (Hb <12g/dL for males, <11g/dL for females)
7. Concomitant or previous conditions that preclude injection of vaccines/infusion of monoclonal antibody and PML in the past
8. History of experimental vaccinations against HIV
9. Previous treatment with chemotherapy (except for chemotherapy injected into skin lesions for Kaposi's sarcoma)
10. Treatment with systemic corticoids or immuno-suppressive agents ongoing or in the previous 12 weeks before randomisation in the trial
11. Received natalizumab or rituximab ever in the past
12. Received a TNF blocker in the past 60 days
13. Administration of an inactivated vaccine within 30 days or a live vaccine within 60 days prior to randomisation
14. Presence of a skin condition or marking that precludes inspection of the injection/infusion site
15. History of cancer (except basal cellular skin carcinoma or Kaposi's sarcoma)
16. History of significant neurological disease, cardiovascular disease (angina, myocardial infarction, transient ischemic attack, stroke); participants with controlled blood pressure are eligible
17. Personal history of clinical autoimmune disease or reactive arthritis or family history of rheumatoid arthritis (parents or siblings)
18. Ongoing diseases including uncontrolled active severe infection, cardiac, pulmonary (excluding mild asthma), thyroid, renal or neurological (peripheral or central) diseases
19. Active or latent tuberculosis (unless prophylaxis in past as per local practice) - (participant must be screened for tuberculosis before starting infusions, according to routine practice)
20. Presence of pathogenic bacteria or parasites in faeces at screening
21. Participating in another biomedical research study within 30 days of randomisation.
22. Known hypersensitivity to any component of the vaccine formulations used in this trial including aminoglycosides and eggs or have severe or multiple allergies to drugs or pharmaceutical agents, or any hypersensitivity to the active substance or to any of the excipients of vedolizumab
23. Liver disease including hepatitis B (surface antigen positive) or hepatitis C (antigen or PCR positive)
24. A clinically significant abnormality on ECG
25. Hypernatraemia or hyperchloraemia
26. History of severe local or general reaction to vaccination defined as

    1. local: extensive, indurated redness and swelling involving most of the arm, not resolving within 72 hours
    2. general: fever >= 39.5oC within 48 hours; anaphylaxis; bronchospasm; laryngeal oedema; collapse; convulsions or encephalopathy within 72 hours
27. Grade 2 or worse routine laboratory parameters (see Appendix 4 for definitions). Hyperbilirubinaemia to be considered an exclusion criterion only when confirmed to be conjugated bilirubinaemia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-02-20 (Actual); Primary Completion 2019-07-11 (Actual); Study Completion 2019-07-11 (Actual)

PRIMARY OUTCOMES:
Efficacy: Time from treatment interruption to the earliest of reaching HIV RNA ≥ 10,000 copies/ml or resuming antiretroviral therapy for any reason over a period of 24 weeks. | Time from treatment interruption (scheduled for 12 weeks after completing the immunisation schedule) to the earliest of reaching HIV RNA ≥ 10,000 copies/ml or resuming antiretroviral therapy for any reason over a period of 24 weeks.
Safety: A clinical decision to discontinue the regimen for an adverse event that is considered related to product | From randomisation

SECONDARY OUTCOMES:
Grade 3 and worse solicited clinical and laboratory adverse events | From randomisation to study completion, about 60 weeks.
Any event leading to interruption in the vaccine schedule | From randomisation to study completion, about 60 weeks.
Any event that results in resuming treatment during the ATI | From randomisation to study completion, about 60 weeks.
Serious Adverse Events | From randomisation to 30 days after the last protocol visit
Other clinical and laboratory adverse events | From randomisation to study completion, about 60 weeks.
Time to VL suppression after restarting ART | From randomisation to VL suppression after restarting ART

OTHER OUTCOMES:
Secondary Immunological Outcomes | From randomisation
  Response rate, magnitude and polyfunctionality of vaccine induced CD4 and CD8 T-cell responses.
Secondary Virological efficacy outcome measures | From randomisation
  Level of HIV total DNA and Cell Associated (CA) HIV RNA Quantification

CONTACTS AND LOCATIONS:
Overall Officials: Yves Levy, MD, Study Director — Institut National de la Santé Et de la Recherche Médicale, France
Locations (2):
- CHUV, Lausanne, Switzerland
- Chelsea & Westminster Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No